CLINICAL TRIAL: NCT02506920
Title: Gender Dependent Difference in Postprandial Lipemia and Glucose Responses After Six Different Fat Tolerance Tests in Young Healthy Subjects
Brief Title: Gender Dependent Difference in Lipemia After 6 x OFTT in Young Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Collaborators: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Finn Friis Lauszus, Senior Consultant, Herning Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Gender and PPL
Record Dates: First submitted 2015-06-26; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Hyperlipidemia
Keywords: Postprandial lipemia; glycemic response
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Pack butter (Active Comparator): Oral fat tolerance test contains: Cream, lactic acid culture, salt. Fat contents in grams: Saturated fat (SFA) 52, monounsaturated fat (MUFA) 19.1, polyunsaturated fat (PUFA) 1.6
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order
- Kjaergaarden blend butter (Active Comparator): Oral fat tolerance test contains:Butter rapeseed oil, lactic acid culture, salt. Fat contents in grams: SFA 37.4, MUFA 27.3, PUFA 1.8
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order
- Blend butter (Active Comparator): Oral fat tolerance test contains: Butter rapeseed oil, lactic acid culture, salt. Fat contents in grams: SFA 23.7, MUFA 23.2, PUFA 7.8
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order
- Fish oil enriched butter (Active Comparator): Oral fat tolerance test contains: Butter rapeseed oil, lactic acid culture, fish oil, salt. Fat contents in grams: SFA 22.6, MUFA 26.9, PUFA 0.7
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order
- Olive oil enriched butter (Active Comparator): Oral fat tolerance test contains: Butter rapeseed oil, olive oil, lactic acid culture, salt. Fat contents in grams: SFA 22.6, MUFA 26.9, PUFA 5.7
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order
- Low saturated fat butter (Active Comparator): Oral fat tolerance test contains: Butter, lactic acid culture, salt. Fat contents in grams: SFA14.9, MUFA16, PUFA 5.6
  Interventions: Dietary Supplement: Six different types of fat in a meal in random order

INTERVENTIONS:
Dietary Supplement: Six different types of fat in a meal in random order — Oral fat tolerance test

SUMMARY:
The investigators wanted to study the postprandial lipemia after six oral fat tolerance test with varying amounts of saturated fat in young healthy subjects.

DETAILED DESCRIPTION:
With six different types of butter added in random order to potatoes the investigators studied postprandial lipemia (PPL), lipoprotein, glucose, and insulin increments for eight hours in 14 young, lean, healthy students, seven of each gender.

The six, isocaloric meals contained 55.1 g carbohydrate, 5.8 g protein, 82.3 g fat, and 4177 kJ. The potatoes, without skin, were boiled in 20 minutes in excess of water with 5 g of salt added, were blended in 4 minutes and served hot. The meals were ingested over 10 minutes, with 250 ml tap water. The following 8 hours the participants stayed at the clinic to watch television, read or take a short walk of 10 minutes.

Blood samples were drawn at -15, 0, 30, 60, 90,120,180,240,300,360, 420 and 480 minutes after the meals and processed after each drawing. After blood collection, plasma was immediately separated by centrifugation at 3000 rpm for 10 minutes at 4°C.

The area under the curve (AUC) were determined for TG, HDL, LDL, total cholesterol, FFA, insulin, and glucose concentrations by the trapezoid method. Multiple regression was performed to adjust for age, gender, meals, and BMI to the variance of postprandial responses. The difference between meals were tested with ANOVA. If p<0.05 in ANOVA, post-hoc-testing with Student-Newman-Keul's test was performed to identify, which meal was significantly different from the other, and to minimize the risk of error by multiple testing.

ELIGIBILITY:
Inclusion Criteria:

* Accept healthy volunteers

Exclusion Criteria:

* hypercholesterolemia,
* hypertension,
* abuse of drugs or alcohol,
* known kidney, liver, heart and metabolic disease
* hormonal therapies including oral contraceptives

Ages: 22 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 1997-01; Primary Completion 1997-04 (Actual); Study Completion 1997-12 (Actual)

PRIMARY OUTCOMES:
Postprandial cholesterol | Eight hours
  Cholesterols measured in milli mol per liter
Postprandial free fatty acids | Eight hours
  Free fatty acids measured in micro equivalents per liter

SECONDARY OUTCOMES:
Postprandial glucose | Eight hours
  Glucose measured in milli mol per liter
postprandial insulin | Eight hours
  Insulin measured in pico mol per liter

CONTACTS AND LOCATIONS:
Overall Officials: Ole W Rasmussen, DrMedScie, Principal Investigator — Associate Professor, Kolding Hospital, Denmark

REFERENCES:
- [Background] Astrup A, Dyerberg J, Elwood P, Hermansen K, Hu FB, Jakobsen MU, Kok FJ, Krauss RM, Lecerf JM, LeGrand P, Nestel P, Riserus U, Sanders T, Sinclair A, Stender S, Tholstrup T, Willett WC. The role of reducing intakes of saturated fat in the prevention of cardiovascular disease: where does the evidence stand in 2010? Am J Clin Nutr. 2011 Apr;93(4):684-8. doi: 10.3945/ajcn.110.004622. Epub 2011 Jan 26. PMID 21270379
- [Background] Ryan MF, O'Grada CM, Morris C, Segurado R, Walsh MC, Gibney ER, Brennan L, Roche HM, Gibney MJ. Within-person variation in the postprandial lipemic response of healthy adults. Am J Clin Nutr. 2013 Feb;97(2):261-7. doi: 10.3945/ajcn.112.047936. Epub 2013 Jan 2. PMID 23283501
- [Background] Knuth ND, Remias DB, Horowitz JF. Adding carbohydrate to a high-fat meal blunts postprandial lipemia in women and reduces meal-derived fatty acids in systemic circulation. Appl Physiol Nutr Metab. 2008 Apr;33(2):315-25. doi: 10.1139/H07-190. PMID 18347687
- [Background] Tentor J, Harada LM, Nakamura RT, Gidlund M, Castilho LN, Cotta de Faria E. Sex-dependent variables in the modulation of postalimentary lipemia. Nutrition. 2006 Jan;22(1):9-15. doi: 10.1016/j.nut.2005.05.004. Epub 2005 Oct 12. PMID 16226013